CLINICAL TRIAL: NCT00301418
Title: Phase I/II Trial of Oral Erlotinib (Tarceva, OSI-774) for Treatment of Relapsed/Refractory Glioblastoma Multiforme and Anaplastic Astrocytoma
Brief Title: Oral Tarceva Study for Recurrent/Residual Glioblastoma Multiforme and Anaplastic Astrocytoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, John A. Boockvar, Professor, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 501007705
Record Dates: First submitted 2006-03-09; First posted 2006-03-10 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-01

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma
Keywords: Glioblastoma Multiforme; Anaplastic Astrocytoma; High Grade Glial Neoplasms; Brain Tumor
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Brain Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tarceva (Erlotinib) (Experimental)
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Tarceva®: Will be given at a starting dose of 150mg QD dose for the first cycle which is 28 days. This will be followed by 14 days of 100mg PO on a bid schedule and 150mg PO on a bid schedule for the final 14 days of the second cycle. Assuming no dose limiting toxicity, 150 mg PO tid will be continued for up to 10 more cycles. This is an outpatient regimen, in which the drug is admininistered orally. Tumor response will be assessed after every 2nd treatment cycle. Patients may receive a maximum of 12 cycles of treatment under this research protocol.
  Other Names: Tarceva; OSI-774

SUMMARY:
This study will offer a safe treatment for patients with relapsing recurring glioblastoma (GBM) or anaplastic astrocytoma (AA). The trial will test the hypothesis that Erlotinib (Tarceva, OSI-774) can be safely used up to a dose of 150 mg two times a day for 12 months to ultimately enhance survival of patients with relapsed/refractory GBM/AA. Correlation of response to Tarceva with particular genetic alterations including epidermal growth factor receptor variant type III (EGFRvIII) amplification and phosphatase and tensin homolog (mutated in multiple advanced cancers 1) (PTEN) loss will be studied.

DETAILED DESCRIPTION:
The high-grade malignant brain tumors, glioblastoma multiforme (GBM) and anaplastic astrocytoma (AA), comprise the majority of all primary brain tumors in adults. This group of tumors also exhibits the most aggressive behavior, resulting in median overall survival durations of only 9-12 months for GBM, and 3-4 years for AA, from initial diagnosis, despite multimodal treatment approaches. Initial therapy consists of either surgical resection, external beam radiation or both. The role of adjuvant or concomitant chemotherapy in the initial therapy of GBM and AA has not, as yet, been clearly defined. Since most of these patients experience a recurrence after first-line therapy, improvements in both first-line and salvage therapy are critical to enhancing quality-of-life and prolonging survival. In August 2003, the U.S. Food and Drug Administration (FDA) granted orphan drug status for Erlotinib in patients with malignant glioma. Erlotinib (OSI-774) has been shown to be active in a range of tumors including GBM, AA and non small cell lung cancer. Because of the promising results in preliminary studies of Erlotinib and because of significant experience with the safety of the dosages proposed in this study, this study will offer a safe adjuvant treatment for patients with relapsing recurring glioblastoma or anaplastic astrocytoma. Therefore, this phase I/II clinical research trial will test the hypothesis that Erlotinib can be safely used up to a dose of 150 mg bid for 12 cycles to ultimately enhance survival of patients with relapsed/refractory GBM/AA with particular genetic alterations including EGFRvIII amplification and PTEN loss.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of ≥ 18 years of age.
* Patients with a documented histologic diagnosis of relapsed or refractory glioblastoma multiforme (GBM), anaplastic astrocytoma (AA) or anaplastic mixed oligoastrocytoma (AOA). All patients will have samples of their tissue evaluated for EGFRvIII overexpression and PTEN loss.
* Patients with a histologically confirmed low grade brain tumor who relapse with an enhancing tumor on magnetic resonance imaging (MRI) can be evaluated for toxicity only.
* Patients must have at least one confirmed and evaluable tumor site.*

  *A confirmed tumor site is one which is biopsy-proven. NOTE: Radiographic procedures (e.g., Gd-enhanced MRI or computed tomography [CT] scans) documenting existing lesions must have been performed within three weeks of treatment on this research study.
* Patients must have a Karnofsky performance status ≥ 60% (or the equivalent Eastern Cooperative Oncology Group [ECOG] level of 0-2) and an expected survival of ≥ three months.
* No chemotherapy for six weeks prior to treatment under this research protocol and no external beam radiation for eight weeks prior to treatment under this research protocol.
* Patients must have adequate hematologic reserve with WBC ≥ 3000/mm3, absolute neutrophils ≥ 1500/mm3 and platelets ≥ 100,000/mm3. Patients who are on Coumadin must have a platelet count of ≥ 150,000/mm3
* Pre-enrollment chemistry parameters must show: bilirubin < 1.5X the institutional upper limit of normal (IUNL); AST or ALT < 2.5X IUNL and creatinine < 1.5X IUNL.
* Pre-enrollment coagulation parameters (PT and PTT) must be ≤ 1.5X the IUNL.
* Concomitant Medications:

  * Growth factor(s): Must not have received within 1 week of entry onto this study.
  * Steroids: Systemic corticosteroid therapy is permissible in patients with centrail nervous system (CNS) tumors for treatment of increased intracranial pressure or symptomatic tumor edema. Patients with CNS tumors who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to study entry.
  * Study Specific: Patients on enzyme-inducing anticonvulsants will be changed to non-enzyme inducing anticonvulsants or will not be allowed on this study. Patients receiving proton pump inhibitor or H2 blockers will not be allowed on study. Patients taking antacids will be allowed on study although they should not take the antacid for two hours before or two hours after taking erlotinib.
* Patients must agree to use a medically effective method of contraception during and for a period of three months after the treatment period. A pregnancy test will be performed on each premenopausal female of childbearing potential immediately prior to entry into the research study.
* Patients should not have received a CYP3A4 inhibitor within 1 week of study entry and should not have received a CYP3A4 inducer within 4 weeks of study entry.
* Patients should not have received proton-pump inhibitors within 5 days of study entry or H2 blockers within 2 days of study entry.
* Patients on steroids must receive prophylaxis for Pneumocystis carinii pneumonia (PCP) with Bactrim, unless they have a history of allergy to sulfa drugs.
* Patients must be able to understand and give written informed consent. Informed consent must be obtained at the time of patient screening.

Exclusion Criteria:

* Previous treatment with Tarceva®.
* Women who are pregnant or lactating.
* Women of childbearing potential and fertile men will be informed as to the potential risk of procreation while participating in this research trial and will be advised that they must use effective contraception during and for a period of three months after the treatment period.
* Patients with significant intercurrent medical or psychiatric conditions that would place them at increased risk or affect their ability to receive or comply with treatment or post-treatment clinical monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Boockvar, M.D., Principal Investigator — Feinstein Institute for Medical Research
Locations (1):
- Lenox Hill Brain Tumor Center, New York, New York, United States

REFERENCES:
- [Background] Mellinghoff IK, Wang MY, Vivanco I, Haas-Kogan DA, Zhu S, Dia EQ, Lu KV, Yoshimoto K, Huang JH, Chute DJ, Riggs BL, Horvath S, Liau LM, Cavenee WK, Rao PN, Beroukhim R, Peck TC, Lee JC, Sellers WR, Stokoe D, Prados M, Cloughesy TF, Sawyers CL, Mischel PS. Molecular determinants of the response of glioblastomas to EGFR kinase inhibitors. N Engl J Med. 2005 Nov 10;353(19):2012-24. doi: 10.1056/NEJMoa051918. PMID 16282176

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tarceva (Erlotinib)
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tarceva (Erlotinib)
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Safety of Twice a Day Oral 150 mg Erlotinib Dosing
Description: Greater than or equal to Grade 2 Adverse Event
Time Frame: duration of the trial
Measure: Number; unit: participants
Arm/Group | Tarceva (Erlotinib)
Number analyzed (Participants) | 11
participants | 9

2. Secondary Outcome: 6-month Progression Free Survival (PFS)
Time Frame: Duration of the trial
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tarceva (Erlotinib)
Number analyzed (Participants) | 11
days | 56 [35.9 to 114.5]

3. Secondary Outcome: Overall Survival (OS)
Time Frame: Duration of the trial
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tarceva (Erlotinib)
Number analyzed (Participants) | 11
days | 167 [98.2 to 227.7]

ADVERSE EVENTS:
Arm/Group | Tarceva (Erlotinib)
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 9/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tarceva (Erlotinib) (N=11)
Rash (Skin and subcutaneous tissue disorders) | 9
Diarrhea (Gastrointestinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes